CLINICAL TRIAL: NCT04234295
Title: Investigating the Effect of Obesity on Eosinophil Recruitment in Human Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elena Anna (Eleanna) De Filippis, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-003803
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Obese; Healthy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lean, Healthy Controls (Active Comparator): Subjects with a body mass index (BMI) of 25 or less will have a fat tissue biopsy collected
  Interventions: Procedure: Fat Tissue Biopsy
- Obese, Non-Diabetic (Experimental): Subject with a BMI between 30 and 50 kg/m2 will have fat tissue biopsy collected
  Interventions: Procedure: Fat Tissue Biopsy

INTERVENTIONS:
Procedure: Fat Tissue Biopsy — If subjects are scheduled for a surgical procedure a fat sample will be collected during the beginning of the surgery. If subjects are not scheduled for a surgical procedure, a small sample of subcutaneous (superficial) fat tissue from subjects abdomen area will be collected.

SUMMARY:
Researchers are trying to better understand the relationship between inflammation in adipose tissue (AT) and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 30-50 years
* Non-smokers
* Lean subjects with a BMI of 25 or less, gender specific normal body fat,
* Obese, non-diabetic subjects with a BMI between 30 and 50 and taking no medications affecting glucose metabolism or lipid metabolism
* subjects scheduled for an elective laparoscopic or laparotomy abdominal surgery

Exclusion Criteria:

* Receiving corticosteroid therapy or have a history of asthma, COPD or atopic syndrome
* taking any biologic treatment for any autoimmune disorder
* Taking any leukotriene receptor antagonist acting medications (ex. Montelukast)
* smoking

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Number of eosinophils in adipose tissue | baseline
  eosinophil number will be measured by flow cytometry in subcutaneous (superficial) adipose tissue

SECONDARY OUTCOMES:
Correlation between eosinophil content and body mass index (BMI) | baseline
  Measured as a linear regression between BMI (defined as the weight in Kg/height in square m; kg/m2) and eosinophil number in the fat

OTHER OUTCOMES:
Quantification of the difference in gene methylation in eosinophils from lean and obese subjects | baseline
  Gene methylation of eosinophils will be quantified in samples derived from lean and obese fat biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Elena De Filippis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez JD, Li T, Ghannam H, Rau CM, Masuda MY, Madura JA 2nd, Jacobsen EA, De Filippis E. Linking adipose tissue eosinophils, IL-4, and leptin in human obesity and insulin resistance. JCI Insight. 2024 Feb 8;9(3):e170772. doi: 10.1172/jci.insight.170772. PMID 38206766
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials